CLINICAL TRIAL: NCT04692077
Title: Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV Among Adolescent Males - A Sub-study of HPTN 083
Brief Title: Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV Among Adolescent Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 083-01; 38654 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2020-12-22; First posted 2020-12-31 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
Keywords: Pre-Exposure Prophylaxis; PrEP
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Tenofovir; Emtricitabine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB LA (Experimental): In Step 1, participants will receive one CAB tablet orally every day for 5 weeks. In Step 2, participants will receive an intramuscular (IM) injection of CAB LA at Weeks 5, 9, 17, 25, and 33. In Step 3, participants will receive a TDF/FTC tablet orally every day for 48 weeks or may be offered the opportunity to join an open label CAB study instead, if such a study is being implemented in their area at the time.
  Interventions: Drug: Cabotegravir (CAB) tablet; Drug: CAB LA; Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) tablet

INTERVENTIONS:
Drug: Cabotegravir (CAB) tablet — 30 mg tablets
Drug: CAB LA — Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter.
Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) tablet — 300 mg/200 mg fixed-dose combination tablets

SUMMARY:
This study will establish the minimum safety, tolerability and acceptability data needed to support the use of cabotegravir long-acting injection (CAB LA) in an adolescent population, potentially transforming the field of HIV prevention for young people.

DETAILED DESCRIPTION:
The purpose of this study is to establish the minimum safety, tolerability and acceptability data needed to support the use of cabotegravir long-acting injection (CAB LA) in an adolescent population, potentially transforming the field of HIV prevention for young people.

This study will enroll healthy, HIV-uninfected adolescents assigned male at birth, including men who have sex with men (MSM), transgender women (TGW), and gender non-conforming people. The total participant commitment for the entire study is approximately 1.5 years.

This study will take place in three steps. In Step 1, participants will receive daily oral CAB tablets for 5 weeks. In Step 2, participants will receive a series of five intramuscular (IM) injections of CAB LA, administered at 8-week intervals after a 4-week loading dose (injections at Weeks 5, 9, 17, 25 & 33). A safety visit will follow each injection to ascertain safety data, including injection site reactions. In Step 3, all participants who have received at least one injection will be followed quarterly (every 3 months) for 48 weeks after their last injection. Participants will receive oral TDF/FTC for daily use for 48 weeks or may be provided the opportunity to enroll in a local open label study of CAB, if available.

Participants will attend about 18 study visits throughout the study. Visits may include physical examinations, blood collection, urine collection, rectal and oral pharyngeal swab collection, risk reduction and adherence counseling, and behavioral or acceptability assessments.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth (includes MSM, TGW, and gender non-conforming people)
* At enrollment, aged below 18 years
* At enrollment, body weight ≥ 35 kg (77 lbs.)
* Willing to provide informed consent for the study
* Self-reported sexual activity with a male in the past 12 months
* In general, good health, as evidenced by the following laboratory values

  * Non-reactive/negative HIV test results
  * Absolute neutrophil count > 799 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 11g/dL
  * Calculated creatinine clearance ≥ 60 mL/minute using modified Schwartz equation (≤ grade 2)
  * Alanine aminotransferase (ALT) < 2.0 times the upper limit of normal (ULN) and total bilirubin (Tbili) ≤ 2.5 x ULN
  * Hepatitis B virus (HBV) surface antigen (HBsAg) negative and accepts vaccination
  * Hepatitis C virus (HCV) Antibody negative
* Willing to undergo all required study procedures
* If currently on pre-exposure prophylaxis (PrEP) from a non-study source, willing to stop said PrEP prior to enrollment and agree to switch to oral CAB for the lead-in period and CAB LA injections.

Exclusion Criteria:

* Co-enrollment in any other HIV interventional research study or other concurrent studies which may interfere with this study (as provided by self-report or other available documentation)
* Past or current participation in HIV vaccine trial with exception for participants who can provide documentation of receipt of placebo
* Exclusively had sex with biological females in lifetime
* In the last 6 months (at the time of screening): active or planned use of any substance which would, in the opinion of the site investigator, would hinder study participation (including herbal remedies), as described in the Investigator's Brochure (IB) or listed in the Study Specific Procedures (SSP), and/ or Protocol Section 4.4
* Known history of clinically significant cardiovascular disease, as defined by history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Inflammatory skin conditions that compromise the safety of intramuscular (IM) injections
* Tattoo or other dermatological condition overlying the buttock region that may interfere with interpretation of injection site reactions
* Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy)
* Known history of clinically significant bleeding
* Surgically-placed or injected buttock implants or fillers, per self-report. Contact the CMC for guidance regarding questions about individual cases
* A history of seizure disorder, per self-report
* Medical, social, or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or the safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* Plans to move out of the geographic area within the next 18 months or otherwise unable to participate in study visits, according to the site investigator.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Assigned male at birth (includes MSM, TGW, and gender non-conforming people)
Enrollment: 9 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — Stroger Hospital of Cook County; Lynda Stranix-Chibanda, MBChB, MMED, Study Chair — University of Zimbabwe College of Health Sciences
Locations (4):
- United States (4):
  - University of Colorado Denver ATN CRS, Aurora, Colorado
  - John H. Stroger Jr. Hosp. of Cook County ATN CRS, Chicago, Illinois
  - The Fenway Institute ATN CRS, Boston, Massachusetts
  - St. Jude Children's Research Hosp. ATN CRS, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study will be targeted towards at-risk, sexually active adolescent populations of MSM in the US. Enrollment will occur over approximately 18 months.
Pre-assignment Details: A total of 9 participants were eligible and enrolled. The Study has 3 steps, Oral CAB, Injection CAB LA and the Follow-up of Injection CAB with use of TDF/FTC, Truvada® for daily use or continued CAB injections for 48 weeks.
  One participant terminated before the end of Step 2 "Withdrawal by Subject". Of the 8 remaining participants, one participant "Scheduled exit visit/end of study" prior to the start of Step 3. Within Step 3, one participant switched from TDF/FTC to Injection CAB LA.
Groups:
- Cabotegravir Long Acting: In Step 1, participants will receive one CAB tablet orally every day for 5 weeks. In Step 2, participants will receive an intramuscular (IM) injection of CAB LA at Weeks 5, 9, 17, 25, and 33. In Step 3, participants will receive a TDF/FTC tablet orally every day for 48 weeks or may be offered the opportunity to join an open label CAB study instead, if such a study is being implemented in their area at the time.
  Cabotegravir (CAB) tablet: 30 mg tablets
  CAB LA: Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter.
  Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) tablet: 300 mg/200 mg fixed-dose combination tablets
Period: Cabotegravir Long Acting Oral Phase
Arm/Group | Cabotegravir Long Acting
Started | 9
Completed | 9
Not Completed | 0
Period: Cabotegravir Long Acting Injection Phase
Arm/Group | Cabotegravir Long Acting
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Step 3 Follow-up Phase
Arm/Group | Cabotegravir Long Acting
Started | 8
CAB LA Injection (Participants who elected to receive intramuscular (IM) cabotegravir (CAB LA) injections during Step 3 follow-up. This regimen consists of 3 mL (600 mg) injections administered every 8 weeks for up to 48 weeks after their final injection in Step 2, with injections given at weeks +8, +16, +24, +32, +40, and +48.) | 5
Tenofovir/Emtricitabine (Participants who elected to receive daily oral Tenofovir/Emtricitabine (TDF/FTC, Truvada®) during Step 3 follow-up. This regimen consists of a 300 mg/200 mg tablet administered daily for up to 48 weeks after their final injection in Step 2, starting at the +8 week visit (then followed at weeks +12, +24, +36, and +48). Participants in Step 3 are permitted to switch from TDF/FTC to CAB LA if desired. One participant did switch from TDF/FTC to CAB LA during Step 3 follow-up.) | 3
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes all enrolled participants.
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (0.7)
Age, Customized [Count of Participants; unit: Participants]
  12-15 years old | 1
  16-17 years old | 8
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-reported Gender Identity
  Participants
    Female | 1
    Gender Nonconforming/Gender Variant | 1
    Male | 6
    Self-Identify | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Age Standardized BMI z-score Classification [Count of Participants; unit: Participants] — Measure Description: Based on age in months. Final z-scores calculated using World Health Organization (WHO) tool
  (https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age).
  Categories allocated according to the following z-scores:
  Obesity: > +2; Overweight: > +1 and <= +2; Normal: > -2 and <= +1; Thinness: > -3 and<= -2; Severe thinness: <= -3.
  Participants
    Obese | 2
    Overweight | 1
    Normal | 6
    Thinness | 0
    Severe thinness | 0
Do you have a regular place or home where you stay and store your things? [Count of Participants; unit: Participants]
  Yes | 9
  No | 0
In the past 6 months, how frequently did you worry that your household would not have enough food? [Count of Participants; unit: Participants]
  Never worried | 8
  Sometimes worried | 0
  Often worried | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Proportion of Participants Experiencing Any Grade 2 or Higher Clinical Adverse Events (AEs) and Laboratory Abnormalities Among Participants Who Receive at Least One Injection of CAB LA.
Description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities (reported as adverse events) from the first injection visit to 8 weeks after the last Step 2 injection visit, or Week 41, whichever comes first.
Time Frame: Measured through participant's first injection visit up to 8 weeks after the last Step 2 injection visit or Week 41, whichever comes first.
Population: Includes enrolled participants who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Groups:
- Cabotegravir Long Acting: Injectable cabotegravir 3 mL (600 mg) intramuscular (IM) injection
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants | 8
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 88.9, 95% CI 2-sided [51.8 to 99.7]; Exact 95% Confidence Interval for Proportion for Participants who Reported Grade 2 and Above AEs

2. Primary Outcome: Tolerability Endpoint: Proportion of Participants Who Receive at Least 1 Injection and Who Discontinue Receiving Injections Prior to the Full Course of Injections Due to Intolerability of Injection, Frequency of Injections or Burden of Study Procedures.
Description: Number and percent of participants who receive at least 1 injection and who discontinue receiving injections prior to the full course of injections due to intolerability of injection or burden of study procedures. Reasons for intolerability may include:
  1. Injection site reaction
  2. Burden of study procedure
     1. Participant refused further participation
     2. Participant is unwilling or unable to comply with required study procedures
     3. Participant refused further study product use
     4. Participant unable to adhere to visit schedule
Time Frame: as for outcome 1
Population: Includes all enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants
  Number of participants who received at least 1 injection of CAB LA | 9
  Number of participants who reported any injection site reaction (ISR) | 5
  Number of participants who have reported any Grade 2 (moderate) or above ISR | 3
  Participants who Discontinued Early due to Intolerability of Injection or Burden of Study Procedure | 1
  Number of participants who completed all scheduled injections | 8
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 11.1, 95% CI 2-sided [0.3 to 48.3]; Exact 95% Confidence Interval for Proportion for Participants who Discontinued Early due to Intolerability of Injection or Burden of Study Procedures

3. Primary Outcome: Acceptability Endpoint: Proportion of Participants Who Complete All Scheduled Injections and Proportion of Participants Who Receive at Least One Injection Whom Would Consider Using CAB LA for HIV Prevention in the Future.
Description: Definition of completing all scheduled injections for participants who are confirmed HIV positive or discontinue product due to the following reasons:
  * Death
  * Early study closure
  * HBV infection
  During Step 2:
  Both enrolled and injection populations: completed all injections whose target window closed prior to death/seroconversion/product discontinuation date
Time Frame: as for outcome 1
Population: Includes all enrolled participants and all enrolled participants who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants
  Participant who received at least one injection among all enrolled participants | 9
  Participants with acceptability endpoint at the end of Step 2 | 6
  Participants who received at least one injection and preferred injectable PrEP at the end of Step 2 | 4
  If you wanted to protect yourself from HIV: Prefer not using a product | 0
  If you wanted to protect yourself from HIV: Condoms only | 1
  If you wanted to protect yourself from HIV: Oral PrEP pills only | 0
  If you wanted to protect yourself from HIV: Injectable PrEP only | 0
  If you wanted to protect yourself from HIV: Condoms and oral PrEP pills together | 1
  If you wanted to protect yourself from HIV: Condoms and injectable PrEP together | 4
  If you wanted to protect yourself from HIV: Prefer not to answer | 0
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 66.7, 95% CI 2-sided [22.3 to 95.7]; Exact 95% confidence interval for proportion for Participants who received at least one injection and preferred injectable PrEP at end of step 2

4. Secondary Outcome: Count of Participant-study Visits Above the Protein-adjusted Inhibitor Concentration (90%; PA-IC90)
Description: CAB drug concentrations will be measured in plasma to generate CAB-LA concentration-time profiles among study participants. Measurements will occur at study visits during the injection phase of the study as well as during the pharmacologic "tail" phase. Count of participants for injection visits in which a participant remains above the 1x (0.166 mcg/mL), 4x (0.664 mcg/mL) and 8x (1.33 mcg/mL) PA-IC90.Concentrations above the 3 PA-IC90 are associated with rectal protection in a non-human primate study, and concentrations above the 8x PA-IC90 are expected to be associated with protection in humans.
Time Frame: Measured from the participant's first injection visit up to 8 weeks after the last Step 2 injection visit or Week 41
Population: Includes enrolled participants who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants
  Injection 1: <1x PA-IC90 | 1
  Injection 1: >=1x - <4x PA-IC90 | 0
  Injection 1: >=4x - <8x PA-IC90 | 0
  Injection 1: >=8x PA-IC90 | 8
  Injection 2: <1x PA-IC90 | 0
  Injection 2: >=1x - <4x PA-IC90 | 1
  Injection 2: >=4x - <8x PA-IC90 | 2
  Injection 2: >=8x PA-IC90 | 6
  Injection 3: number analyzed (Participants) | 8
  Injection 3: <1x PA-IC90 | 0
  Injection 3: >=1x - <4x PA-IC90 | 1
  Injection 3: >=4x - <8x PA-IC90 | 0
  Injection 3: >=8x PA-IC90 | 7
  Injection 4: number analyzed (Participants) | 8
  Injection 4: <1x PA-IC90 | 0
  Injection 4: >=1x - <4x PA-IC90 | 0
  Injection 4: >=4x - <8x PA-IC90 | 2
  Injection 4: >=8x PA-IC90 | 6
  Injection 5: number analyzed (Participants) | 7
  Injection 5: <1x PA-IC90 | 0
  Injection 5: >=1x - <4x PA-IC90 | 0
  Injection 5: >=4x - <8x PA-IC90 | 1
  Injection 5: >=8x PA-IC90 | 6
  Step 3 +8 weeks: number analyzed (Participants) | 7
  Step 3 +8 weeks: <1x PA-IC90 | 0
  Step 3 +8 weeks: >=1x - <4x PA-IC90 | 0
  Step 3 +8 weeks: >=4x - <8x PA-IC90 | 0
  Step 3 +8 weeks: >=8x PA-IC90 | 7

5. Secondary Outcome: Measure Study Product Concentrations in Enrolled Participants With HPTN Laboratory Center (LC) Confirmed HIV Infection Throughout Study.
Description: For infections occurring prior to (or on the first day of) Step 3, we will include visit level plasma CAB concentrations, for individual seroconverters. For infections occurring after the start of Step 3, we will include visit level plasma CAB concentrations as well as concentrations of TFV and TFV-DP (if applicable).
Time Frame: Measured through seroconverter's first Oral visit up through end of study participation (step1, 2, 3)
Population: All enrolled participants who became HIV infected during the study (Step 1, 2 or 3).
  Serum concentrations were not collected for this measure because no participants had HPTN Laboratory Center (LC) Confirmed HIV Infection at enrollment or during Steps 1,2, and 3.
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 0

6. Secondary Outcome: Count and Percentage of Participants Experiencing Grade 2 or Higher Clinical AEs and LaboratoryAbnormalities in the Oral Phase and the Aggregate Oral and Injection Phases
Description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities from:
  1. enrollment to week 5 (oral phase (step 1), including interim visits).
  2. enrollment to 8 weeks following the last injection received (aggregate over oral + injection phases (step 1-step 2) including interim visits)
Time Frame: Measured through participant's first oral visit up to 8 weeks after the last Step 2 injection visit or Week 41, whichever comes first.
Population: Includes enrolled participants who began step 1 (oral phase).
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants
  Number of participants with Grade 2 or Higher AEs in Oral Phase | 3
  Number of participants with Grade 2 or Higher AEs in Oral and Injection Phase | 8

7. Secondary Outcome: Proportion of Participants Receiving One or More Injections Who Experience Grade 2 or Higher Clinical AEs and Laboratory Abnormalities From Initial Injection to 36 Weeks Later.
Description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities from the first injection visit to approximately 36 weeks later regardless of whether participants received all 5 injections.
Time Frame: as for outcome 1
Population: Includes enrolled participants who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants | 8
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 88.9, 95% CI 2-sided [51.8 to 99.7]; The Exact 95% Confidence Interval for Proportion for Number of Participants with Grade 2 or above AEs during Injection Phase

8. Secondary Outcome: Proportion of Injection Visits That Occurred "On-time".
Description: Number and percentage of injections given, using the number of injections expected as the denominator. while the number and percent of injection visits (up to 5 per participant) that occur "on-time", using the number of injections given as the denominator. This will be presented along with the total number and percent of injections given, among all intended injections (i.e. 5 injections per participant).
  Those who have been terminated, are HIV infected, or have permanently discontinued study products at the time of visit will be excluded from the number of expected injections.
Time Frame: Measured through participant's last step 2 injection.
Population: Includes enrolled participants who receive at least one injection of CAB LA.
  By the end of step 2, just 1/8 participants missed their last injection but continued with the study and received a step 3 injection. This participant was counted as having 100% of injections completed with 5 injections. For this analysis, through the end of Step 2, technically 1 less injection was given in this case.
Measure: Number; unit: Number of Injections given
Units Other Than Participants: Number of Injections Expected
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Number analyzed (Number of Injections Expected) | 41
Number of Injections given
  Number of injections given | 40
  Number of injections given on-time: number analyzed (Number of Injections Expected) | 40
  Number of injections given on-time | 32
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 88.9, 95% CI 2-sided [51.8 to 99.7]; Exact 95% Confidence Interval for Proportion for Participants who Completed All Scheduled Injections among those who received at least one Injection

9. Secondary Outcome: Change From Enrollment of Self-reported Sexual Behavior (Number of Sexual Partners) During the Study Period
Description: Counts of sexual partners will be summarized (mean and sd) at enrollment and each regular Step 1 and Step 2 follow-up visit (W4, W5, W9, W17, W25, W33).
Time Frame: Measured through participant's first oral visit up to last Step 2 injection visit.
Population: Includes all enrolled participants:
  For each visits: analysis population includes participants with non-missing value.
  For the difference between 2 visits: analysis population only includes participants with non-missing values for both visits. .
Measure: Mean (Standard Deviation); unit: Number of Sexual Partners
Groups:
- Cabotegravir Long Acting: In Step 1, participants will receive one CAB tablet orally every day for 5 weeks.
  In Step 2, participants will receive an intramuscular (IM) injection of CAB LA at Weeks 5, 9, 17, 25, and 33.
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Number of Sexual Partners
  Enrollment | 0 (0.4)
  Week 4: number analyzed (Participants) | 8
  Week 4 | 0 (0.5)
  Week 4: Change from previous visit: number analyzed (Participants) | 8
  Week 4: Change from previous visit | 0 (0.0)
  Week 4: Change from baseline: number analyzed (Participants) | 8
  Week 4: Change from baseline | 0 (0.0)
  Week 5: number analyzed (Participants) | 8
  Week 5 | 0 (0.7)
  Week 5: Change from previous visit: number analyzed (Participants) | 8
  Week 5: Change from previous visit | 0 (0.4)
  Week 5: Change from baseline: number analyzed (Participants) | 8
  Week 5: Change from baseline | 0 (0.4)
  Week 9: number analyzed (Participants) | 8
  Week 9 | 0 (0.4)
  Week 9: Change from previous visit: number analyzed (Participants) | 8
  Week 9: Change from previous visit | 0 (0.7)
  Week 9: Change from baseline: number analyzed (Participants) | 8
  Week 9: Change from baseline | 0 (0.4)
  Week 17: number analyzed (Participants) | 8
  Week 17 | 0 (0.4)
  Week 17: Change from previous visit: number analyzed (Participants) | 7
  Week 17: Change from previous visit | 0 (0.0)
  Week 17: Change from baseline: number analyzed (Participants) | 8
  Week 17: Change from baseline | 0 (0.4)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 0 (0.4)
  Week 25: Change from previous visit: number analyzed (Participants) | 8
  Week 25: Change from previous visit | 0 (0.0)
  Week 25: Change from baseline: number analyzed (Participants) | 8
  Week 25: Change from baseline | 0 (0.4)
  Week 33: number analyzed (Participants) | 7
  Week 33 | 0 (0.4)
  Week 33: Change from previous visit: number analyzed (Participants) | 7
  Week 33: Change from previous visit | 0 (0.0)
  Week 33: Change from baseline: number analyzed (Participants) | 7
  Week 33: Change from baseline | 0 (0.4)

10. Secondary Outcome: Change From Enrollment of Self-reported Sexual Behavior (Number of Episodes of Anal Intercourse Without a Condom) During the Study Period
Description: Counts of episodes of anal intercourse without a condom will be summarized (mean and sd) at enrollment and each regular Step 1 and Step 2 follow-up visit (W4, W5, W9, W17, W25, W33).
Time Frame: Measured through participant's first oral visit up to the last Step 2 injection visit.
Population: Includes all enrolled participants:
  For each visits: analysis population includes participants with non-missing value.
  For the difference between 2 visits: analysis population only includes participants with non-missing values for both visits.
Measure: Mean (Standard Deviation); unit: Episodes of condomless anal intercourse
Arm/Group | CAB LA
Number analyzed (Participants) | 9
Episodes of condomless anal intercourse
  Enrollment | 1 (1.3)
  Week 4 | 1 (2.3)
  Week 4: Change from previous visit | 0 (1.1)
  Week 4: Change from baseline | 0 (1.1)
  Week 5: number analyzed (Participants) | 8
  Week 5 | 0 (0.7)
  Week 5: Change from previous visit: number analyzed (Participants) | 8
  Week 5: Change from previous visit | -1 (1.8)
  Week 5: Change from baseline: number analyzed (Participants) | 8
  Week 5: Change from baseline | 0 (0.7)
  Week 9: number analyzed (Participants) | 8
  Week 9 | 0 (0.4)
  Week 9: Change from previous visit: number analyzed (Participants) | 8
  Week 9: Change from previous visit | 0 (0.4)
  Week 9: Change from baseline: number analyzed (Participants) | 8
  Week 9: Change from baseline | -1 (1.1)
  Week 17: number analyzed (Participants) | 8
  Week 17 | 0 (1.1)
  Week 17: Change from previous visit: number analyzed (Participants) | 7
  Week 17: Change from previous visit | 0 (0.8)
  Week 17: Change from baseline: number analyzed (Participants) | 8
  Week 17: Change from baseline | 0 (0.5)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 0 (0.7)
  Week 25: Change from previous visit: number analyzed (Participants) | 8
  Week 25: Change from previous visit | 0 (0.4)
  Week 25: Change from baseline: number analyzed (Participants) | 8
  Week 25: Change from baseline | 0 (0.7)
  Week 33: number analyzed (Participants) | 7
  Week 33 | 0 (0.0)
  Week 33: Change from previous visit: number analyzed (Participants) | 7
  Week 33: Change from previous visit | 0 (0.8)
  Week 33: Change from baseline: number analyzed (Participants) | 7
  Week 33: Change from baseline | -1 (1.5)

11. Secondary Outcome: Evaluate Rates of HIV Drug Resistance Among Participants Who Acquire HIV Infection During the Study
Description: Data from steps 1, 2, and 3 will be included. The number of cases of drug resistance will be summarized. All cases of drug resistance among incident HIV infections will be described.
Time Frame: Measured through participant's last study visit, up to approximately 1.5 years after study entry.
Population: Includes all enrolled participants who seroconverted during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 9
Participants
  Number of participants HIV-positive at enrollment | 0
  Number of participants infected | 0
  Number of drug resistant cases | 0

ADVERSE EVENTS:
Time Frame: Measured from participant's first Oral visit up to follow-up 48 weeks Step 3.
Description: SAE, NON SAE, and Mortality are summarized by Steps (Oral, Injection & Follow-up)
Groups:
- Step 1 - CAB LA Oral Phase: A 5-week oral CAB 30 mg QD safety lead-in
- Step 2 - CAB LA Injection Phase: A series of 5 intramuscular (IM) injections of 3 mL (600 mg) cabotegravir administered at 8 week intervals after a 4-week loading dose (injections at weeks 5, 9, 17, 25 & 33)
- Step 3 - CAB LA Injection Follow-up: Participants who elected to receive intramuscular (IM) cabotegravir (CAB LA) injections during Step 3 follow-up. This regimen consists of 3 mL (600 mg) injections administered every 8 weeks for up to 48 weeks after their final injection in Step 2, with injections given at weeks +8, +16, +24, +32, +40, and +48.
- Step 3 - Tenofovir/Emtricitabine Follow-up: Participants who elected to receive daily oral Tenofovir/Emtricitabine (TDF/FTC, Truvada®) during Step 3 follow-up. This regimen consists of a 300 mg/200 mg tablet administered daily for up to 48 weeks after their final injection in Step 2, starting at the +8 week visit (then followed at weeks +12, +24, +36, and +48). Participants in Step 3 are permitted to switch from TDF/FTC to CAB LA if desired.
Arm/Group | Step 1 - CAB LA Oral Phase | Step 2 - CAB LA Injection Phase | Step 3 - CAB LA Injection Follow-up | Step 3 - Tenofovir/Emtricitabine Follow-up
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 1/6 | 0/3
Other Adverse Events (participants affected / at risk) | 8/9 | 9/9 | 5/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step 1 - CAB LA Oral Phase (N=9) | Step 2 - CAB LA Injection Phase (N=9) | Step 3 - CAB LA Injection Follow-up (N=6) | Step 3 - Tenofovir/Emtricitabine Follow-up (N=3)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step 1 - CAB LA Oral Phase (N=9) | Step 2 - CAB LA Injection Phase (N=9) | Step 3 - CAB LA Injection Follow-up (N=6) | Step 3 - Tenofovir/Emtricitabine Follow-up (N=3)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 2 (2) | 4 (5) | 0 (0) | 1 (2)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 3 (3) | 6 (9) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04692077/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT04692077/SAP_002.pdf